CLINICAL TRIAL: NCT04650191
Title: Surfactant Protein Genetic Variants in COVID-19 Infection
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Chintan Gandhi, Assistant Professor, Milton S. Hershey Medical Center
Other Study IDs: 15456
Record Dates: First submitted 2020-11-30; First posted 2020-12-02 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — DNA will be stored for the future studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild COVID-19 infection: Patients with confirmed COVID-19 infection who remained asymptomatic and/or never hospitalized.
  Interventions: Other: Identification of genetic variants
- Moderate COVID-19 infection: Patients with confirmed COVID-19 infection who got admitted in general ward in the hospital.
  Interventions: Other: Identification of genetic variants
- Severe COVID-19 infection: Patients with confirmed COVID-19 infection who got admitted in intensive care unit and/or did not survive.
  Interventions: Other: Identification of genetic variants

INTERVENTIONS:
Other: Identification of genetic variants — DNA will be extracted from whole blood from study subjects

SUMMARY:
Surfactant protein plays important role in innate immunity against respiratory viral infections. However, investigators have shown that the surfactant protein polymorphisms are associated with severity of various pulmonary diseases such as respiratory syncytial virus (RSV), tuberculosis, pediatric acute lung injury. COVID-19 virus gains entry through the respiratory system and responsible for death due to acute respiratory failure. There is a considerable heterogeneity in presentation of COVID-19 infection from asymptomatic patients to severe infection requiring intensive care and some may die. Considering reports of COVID-19 related deaths/severe disease in the same family, it is possible that genetics play an important role in severity of COVID-19 infection. Investigators propose to study the association of surfactant proteins in COVID-19 patients. Key Objectives: a) Characterize genetic markers within the surfactant protein genes in COVID-19 positive patients, b) To determine if there is a correlation between certain genetic markers and the severity of COVID-19 infection which may be used as a prognostic marker, c) To correlate genetic markers with immune studies.

ELIGIBILITY:
Inclusion Criteria:

The major inclusion criteria is a confirmed diagnosis of COVID-19 infection performed on nasopharyngeal secretions by enzyme immunoassay or culture in patients.

Exclusion Criteria:

Patients unable to sign informed consent will be excluded.

Ages: 1 Day to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with positive COVID-19 infection will be enrolled regardless of age and sex after obtaining informed consent.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Correlation of surfactant protein genetic variants with severity of COVID-19 infection | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Milton S. Hershey Medical center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be available to other researchers.